CLINICAL TRIAL: NCT05543265
Title: Bridging the Gap From Postpartum to Primary Care: A Behavioral Science Informed Intervention to Improve Chronic Disease Management Among Postpartum Women
Brief Title: Bridging the Gap From Postpartum to Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Bureau of Economic Research, Inc. (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Mark Clapp, MD MPH, Physician Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022P001723; P30AG034532 (NIH); P30AG064190 (NIH)
Record Dates: First submitted 2022-09-06; First posted 2022-09-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Hypertension in Pregnancy; Diabetes Mellitus; Gestational Diabetes; Obesity; Depressive Disorder; Anxiety Disorders
Keywords: Postpartum Care; Primary Care; Care Transitions
MeSH Terms: conditions — Hypertension; Hypertension, Pregnancy-Induced; Diabetes Mellitus; Diabetes, Gestational; Obesity; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine postpartum care
- Facilitated Transition (Experimental): Behavioral science informed interventions to assist in the transition from postpartum to primary care providers
  Interventions: Behavioral: Default appointment scheduling; Behavioral: Targeted messaging; Behavioral: Nudge Reminders

INTERVENTIONS:
Behavioral: Default appointment scheduling — Default primary care appointment scheduling
  Arms: Facilitated Transition
Behavioral: Targeted messaging — Patient-specific messages about the importance of postpartum care transition
  Arms: Facilitated Transition
Behavioral: Nudge Reminders — Primary care appointment reminders
  Arms: Facilitated Transition

SUMMARY:
Chronic health conditions affect most older adults. Preventative medicine and risk management strategies, especially when applied earlier in life, are essential to altering the trajectory of a disease and ultimately improving health outcomes. Primary care providers (PCP) often provide most of these services, though younger adults are the least likely to receive primary care. This project leverages a period of high engagement and health activation during an individual's life (pregnancy) to nudge her toward use of primary care after the pregnancy episode. This randomized controlled trial will test the hypothesis that a behavioral science-informed intervention, incorporating defaults and salience, can increase the rates of PCP follow-up within 4 months following a delivery for individual with hypertension, diabetes, obesity. If successful, this intervention could serve as a scalable solution to increase primary care use and preventative health services in a population that currently has low rates of engagement and utilization of these services.

DETAILED DESCRIPTION:
Individuals will be randomized with equal probability into either a treatment or control arm. The intervention combines several features designed to target reasons for low take-up of primary care among postpartum individuals. This project will leverage the potential value of defaults/opt-out, salient information, and reminders to encourage use of primary care. Individuals in both the intervention and control arms will receive information via the study institution's patient portal toward the end of the pregnancy regarding the importance and benefits of primary care in the postpartum year. This information will be similar to, but reinforcing, the information they would receive from their obstetrician about following up with their primary care physician. In addition to this initial message, individuals in the treatment arm will receive the following intervention components, developed based on recent evidence regarding behavioral science approaches to activating health behaviors:

1. Targeted messages about the importance and benefits of primary care
2. Default scheduling into a primary care appointment at approximately 3-4 months after delivery
3. Reminders about the appointment and importance of follow up primary care at 2-4 points during the postpartum period via the patient portal
4. Tailored language in the reminders based on recent evidence from behavioral science about the most effective approaches to increasing take-up. For example, messages will inform the patient that an appointment is being held for them at their doctor.
5. Salient labeling on follow-up appointments
6. Direct PCP messaging about the scheduled follow-up

ELIGIBILITY:
Inclusion Criteria:

* Estimated date of delivery and the following 4-month postpartum outcome assessment window completed prior to study end date
* Currently pregnant or within 2 weeks of delivery
* Have one or more of the following conditions: 1) Chronic hypertension, 2) Hypertensive disorders of pregnancy or risk factors for hypertensive disorders of pregnancy per the USPSTF aspirin prescribing guidelines (e.g., history of pre-eclampsia, kidney disease, multiple gestation, autoimmune disease), 3) Type 1 or 2 diabetes, 4) Gestational diabetes, 5) Obesity (pre-pregnancy body mass index ≥30 kg/m2), 6) Depression or anxiety disorder
* Have a primary care provider listed in the electronic health record (EHR)
* Receive obstetric care at the study institution's outpatient prenatal clinic
* Have access to and be enrolled in the EHR patient portal and consents to be contacted via these modalities
* Able to read/speak English or Spanish language
* Age ≥18 years old
* Not actively known to have or undergoing work-up for fetal demise

Exclusion Criteria:

* No primary care provider listed in the EHR
* Primary language other than English or Spanish
* No access to online patient EHR portal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Clapp, MD, MPH, Principal Investigator — Massachusetts General Hospital; Jessica L Cohen, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delgado A, Liang P, Bender T, Ray A, James KE, Ganguli I, Cohen JL, Clapp MA. Primary Care Utilization Within 1 Year After a Facilitated Postpartum-to-Primary Care Transition. Obstet Gynecol. 2025 Apr 1;145(4):409-416. doi: 10.1097/AOG.0000000000005848. Epub 2025 Feb 13. PMID 40117132
- [Derived] Clapp MA, Ray A, Liang P, James KE, Ganguli I, Cohen JL. Postpartum Primary Care Engagement Using Default Scheduling and Tailored Messaging: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2422500. doi: 10.1001/jamanetworkopen.2024.22500. PMID 39012630
- [Derived] Clapp MA, Ray A, Liang P, James KE, Ganguli I, Cohen J. Increasing Postpartum Primary Care Engagement through Default Scheduling and Tailored Messaging: A Randomized Clinical Trial. medRxiv [Preprint]. 2024 May 1:2024.01.21.24301585. doi: 10.1101/2024.01.21.24301585. PMID 38633772

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Facilitated Transition
Started | 176 | 184
Completed | 173 | 180
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients receiving care at 6 outpatient clinics affiliated with a single hospital in Eastern Massachusetts
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Facilitated Transition | Total
Number analyzed (Participants) | 173 | 180 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (5.0) | 34.2 (4.8) | 34.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 180 | 353
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 37 | 78
  Not Hispanic or Latino | 127 | 139 | 266
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 00 | 0 | 0
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 115 | 127 | 242
  More than one race | 28 | 25 | 53
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 173 | 180 | 353

OUTCOME MEASURES:

1. Primary Outcome: Rate of Primary Care Provider Visit Attendance
Description: Any visit with 1) a primary care provider (e.g., internal medicine, family medicine, pediatrics, gynecology) and 2) receipt of "annual" or "health care maintenance" services OR disease-specific management (diabetes, hypertension, obesity, mental health)
Time Frame: 4 months after the patient's estimated date of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Facilitated Transition
Number analyzed (Participants) | 173 | 180
Participants | 38 | 72
Statistical Analysis 1: Comparison: Control vs Facilitated Transition; Test type: Superiority; p < 0.001, Chi-squared; Mean Difference (Final Values) = 22.0, 95% CI 2-sided [6.4 to 28.8]

2. Secondary Outcome: Rate of Primary Care Provider Visit Attendance
Description: as for outcome 1
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

3. Secondary Outcome: Rate of Visit With a Patient's Assigned Primary Care Provider for Receipt of "Annual" or "Health Care Maintenance" Services OR Disease-specific Management (Diabetes, Hypertension, Obesity, Mental Health)
Description: Health care maintenance visit appointment with the patient's assigned primary care provider
Time Frame: 4 months after the patient's estimated date of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Facilitated Transition
Number analyzed (Participants) | 173 | 180
Participants | 30 | 58

4. Secondary Outcome: Rate of Visit With a Patient's Assigned Primary Care Provider for Receipt of "Annual" or "Health Care Maintenance" Services OR Disease-specific Management (Diabetes, Hypertension, Obesity, Mental Health)
Description: Health care maintenance visit appointment with the patient's assigned primary care provider
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

5. Secondary Outcome: Rate of Visit Unscheduled Health Care Visit/Encounter by the Time of Outcome Assessment
Description: Any visit to a urgent care or emergency room visit
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Visit Unscheduled Health Care Visit/Encounter
Description: Any visit to a urgent care or emergency room visit
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

7. Secondary Outcome: Rate of Contraception Plan Documented by the Time of Outcome Assessment
Description: Contraception plan documented by any provider after delivery
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

8. Secondary Outcome: Rate of Long-acting Contraception Use at Time of Outcome Assessment
Description: Long-acting contraception use (implant, intrauterine device)
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

9. Secondary Outcome: Rate of Long-acting Contraception Use
Description: Long-acting contraception use (implant, intrauterine device)
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

10. Secondary Outcome: Rate of Contraception Plan Documented
Description: Contraception plan documented by any provider after delivery
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

11. Secondary Outcome: Rate of Pregestational Diabetes Screening Among Individuals With Gestational Diabetes
Description: Postpartum diabetes screening among those diagnosed with gestational diabetes
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

12. Secondary Outcome: Rate of Pregestational Diabetes Screening Among Individuals With Gestational Diabetes
Description: Postpartum diabetes screening among those diagnosed with gestational diabetes
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

13. Secondary Outcome: Rate of Weight Counseling Documented in the Health Record Among Those With Obesity
Description: Weight counseling documentation among those with obesity
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

14. Secondary Outcome: Rate of Weight Counseling Documented in the Health Record Among Those With Obesity
Description: Weight counseling documentation among those with obesity
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

15. Secondary Outcome: Rate of Blood Pressure Measurement Documented in the Health Record Among Those With or at Risk for Hypertension
Description: Blood pressure documented in the EHR among those diagnosed within chronic or pregnancy-related hypertension
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

16. Secondary Outcome: Rate of Blood Pressure Measurement Documented in the Health Record Among Those With or at Risk for Hypertension
Description: Blood pressure documented in the EHR among those diagnosed within chronic or pregnancy-related hypertension
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

17. Secondary Outcome: Rate of Mental Health Service Referral or Use Among Individuals With Mood or Anxiety Disorders
Description: Clinical support services (e.g., social work, psychiatry, therapy) for individuals with mood or anxiety disorders
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

18. Secondary Outcome: Rate of Mental Health Service Referral or Use Among Individuals With Mood or Anxiety Disorders
Description: Clinical support services (e.g., social work, psychiatry, therapy) for individuals with mood or anxiety disorders
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

19. Secondary Outcome: Rate of Antidepressant Use Among Individuals With Mood or Anxiety Disorders
Description: New or continued antidepressant prescription use
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

20. Secondary Outcome: Rate of Antidepressant Use Among Individuals With Mood or Anxiety Disorders
Description: New or continued antidepressant prescription use
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

21. Secondary Outcome: Rate of Antihypertensive Use Among Individuals With Hypertension
Description: New or continued antihypertensive medication use among individuals with hypertension
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

22. Secondary Outcome: Rate of Antihypertensive Use Among Individuals With Hypertension
Description: New or continued antihypertensive medication use among individuals with hypertension
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

23. Secondary Outcome: Rate of Medication Use for Glycemic Control Among Individuals With Diabetes
Description: New or continued oral or subcutaneous diabetes medication use control among individuals with diabetes
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

24. Secondary Outcome: Rate of Medication Use for Glycemic Control Among Individuals With Diabetes
Description: New or continued oral or subcutaneous diabetes medication use control among individuals with diabetes
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

25. Secondary Outcome: Rate of Assessment of Glycemic Control Among Individuals With or at Risk for Diabetes
Description: Laboratory glucose screening test among individuals with or at risk for diabetes
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

26. Secondary Outcome: Rate of Assessment of Glycemic Control Among Individuals With or at Risk for Diabetes
Description: Laboratory glucose screening test among individuals with or at risk for diabetes
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

27. Secondary Outcome: Rate of Patient-reported Primary Care Visit Attendance
Description: Primary care provider visit attendance per patient report
Time Frame: 4 months after the patient's estimated date of delivery
Reporting Status: Not Posted

28. Secondary Outcome: Rate of Patient-reported Primary Care Visit Attendance
Description: Primary care provider visit attendance per patient report
Time Frame: 12 months after the patient's estimated date of delivery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | Facilitated Transition
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/180
Other Adverse Events (participants affected / at risk) | 0/173 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT05543265/Prot_SAP_ICF_000.pdf